CLINICAL TRIAL: NCT01309633
Title: Phase II Open-label Study Evaluating Two Loading Regimens of Sunitinib or Bevacizumab Alternating With Cisplatin and Gemcitabine as Systemic Therapy for Locally Advanced or Metastatic Nasopharyngeal Carcinoma (NPC)
Brief Title: Study Evaluating Two Loading Regimens of Sunitinib or Bevacizumab Alternating With Cisplatin and Gemcitabine as Induction Therapy for Locally Advanced Nasopharyngeal Carcinoma (NPC)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National University Hospital, Singapore (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NP01/27/10
Record Dates: First submitted 2011-03-03; First posted 2011-03-07 (Estimated); Last update posted 2019-07-22 (Actual); Status verified 2019-07

CONDITIONS: Nasopharyngeal Carcinoma
Keywords: locally advanced; metastatic
MeSH Terms: conditions — Nasopharyngeal Carcinoma; Neoplasm Metastasis | interventions — Sunitinib; Cisplatin; Gemcitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Arm A (Experimental): 1) Arm A
  Day -6 to Day 0 (total 7 days):
  Sunitinib 12.5mg daily Cycles 1 and 2 - Day 1: IV Gemcitabine 1000mg/m2 + IV Cisplatin 75mg/m2 Day 8: IV Gemcitabine 1000mg/m2 Day 15 to Day 21: Sunitinib 12.5mg daily Cycle 3 - Day 1: IV Gemcitabine 1000mg/m2 + IV Cisplatin 75mg/m2 Day 8: IV Gemcitabine 1000mg/m2
  Interventions: Drug: 12.5mg sunitinib with Cisplatin and Gemcitabine
- Arm B (Experimental): Arm B
  Day -6 to Day 0 (total 7 days):
  Sunitinib 25mg daily Cycles 1 and 2 - Day 1: IV Gemcitabine 1000mg/m2 + IV Cisplatin 75mg/m2 Day 8: IV Gemcitabine 1000mg/m2 Day 15 to Day 21: Sunitinib 25mg daily Cycle 3 - Day 1: IV Gemcitabine 1000mg/m2 + IV Cisplatin 75mg/m2 Day 8: IV Gemcitabine 1000mg/m2
  Interventions: Drug: 25mg Sunitinib alternating with Cisplatin and Gemcitabine
- Arm C (Experimental): Arm C Day -7: IV bevacizumab 7.5mg/kg diluted in normal saline over 30 minutes Day 1: IV Gemcitabine 1000mg/m2 + IV Cisplatin 75mg/m2 Day 8: IV Gemcitabine 1000mg/m2 For locally advanced patients, 3 cycles of treatment will be administered. For metastatic patients, up to 6 cycles would be administered.
  Interventions: Drug: 7.5mg/kg Bevacizumab alternating with Cisplatin and Gemcitabine
- Arm D (Experimental): Arm D Day -7: IV bevacizumab 2.5mg/kg diluted in normal saline over 30 minutes Day 1: IV Gemcitabine 1000mg/m2 + IV Cisplatin 75mg/m2 Day 8: IV Gemcitabine 1000mg/m2 For locally advanced patients, 3 cycles of treatment will be administered. For metastatic patients, up to 6 cycles would be administered
  Interventions: Drug: 2.5mg/kg Bevacizumab alternating with Cisplatin and Gemcitabine

INTERVENTIONS:
Drug: 12.5mg sunitinib with Cisplatin and Gemcitabine — 1) Arm A
  Day -6 to Day 0 (total 7 days):
  Sunitinib 12.5mg daily Cycles 1 and 2 - Day 1: IV Gemcitabine 1000mg/m2 + IV Cisplatin 75mg/m2 Day 8: IV Gemcitabine 1000mg/m2 Day 15 to Day 21: Sunitinib 12.5mg daily Cycle 3 - Day 1: IV Gemcitabine 1000mg/m2 + IV Cisplatin 75mg/m2 Day 8: IV Gemcitabine 1000mg/m2
  Other Names: Arm A
  Arms: Arm A
Drug: 25mg Sunitinib alternating with Cisplatin and Gemcitabine — Arm B
  Day -6 to Day 0 (total 7 days):
  Sunitinib 25mg daily Cycles 1 and 2 - Day 1: IV Gemcitabine 1000mg/m2 + IV Cisplatin 75mg/m2 Day 8: IV Gemcitabine 1000mg/m2 Day 15 to Day 21: Sunitinib 25mg daily Cycle 3 - Day 1: IV Gemcitabine 1000mg/m2 + IV Cisplatin 75mg/m2 Day 8: IV Gemcitabine 1000mg/m2
  Other Names: Arm B
  Arms: Arm B
Drug: 7.5mg/kg Bevacizumab alternating with Cisplatin and Gemcitabine — Day -7: IV bevacizumab 7.5mg/kg diluted in normal saline over 30 minutes Day 1: IV Gemcitabine 1000mg/m2 + IV Cisplatin 75mg/m2 Day 8: IV Gemcitabine 1000mg/m2 For locally advanced patients, 3 cycles of treatment will be administered. For metastatic patients, up to 6 cycles would be administered.
  Other Names: Arm C
  Arms: Arm C
Drug: 2.5mg/kg Bevacizumab alternating with Cisplatin and Gemcitabine — Day -7: IV bevacizumab 2.5mg/kg diluted in normal saline over 30 minutes Day 1: IV Gemcitabine 1000mg/m2 + IV Cisplatin 75mg/m2 Day 8: IV Gemcitabine 1000mg/m2 For locally advanced patients, 3 cycles of treatment will be administered. For metastatic patients, up to 6 cycles would be administered
  Other Names: Arm D
  Arms: Arm D

SUMMARY:
- Hypothesis

We hypothesise that intermittent dosing of the anti-angiogenic RTKI sunitinib or bevacizumab prior to systemic cisplatin and gemcitabine chemotherapy to transiently "normalise" tumour vasculature in patients with locally advanced or metastatic NPC will allow greater efficiency in drug and oxygen delivery, thus potentiating sensitivity to chemotherapy. We hypothesise that a loading dose of sunitinib for 7 days is required to achieve this sensitization effect prior to the first cycle of chemotherapy, and that this effect can subsequently be maintained by a 7 day course of sunitinib prior to each subsequent cycle of chemotherapy. The other hypothesis tested is that bevacizumab 7 days prior to chemotherapy will achieve normalization of tumor vasculature as well, and may induce changes in the tumor microenvironment that is beneficial for antitumour effect.

DETAILED DESCRIPTION:
* Primary objectives

  1. To determine the pathological CR* rate of intermittent sunitinib or bevacizumab administered with combination cisplatin and gemcitabine as systemic therapy for locally advanced or metastatic NPC.
  2. To determine the safety and tolerability of intermittent sunitinib or bevacizumab administered with combination cisplatin and gemcitabine as systemic therapy for locally advanced or metastatic NPC.
* Secondary objectives

  1. To determine the clinical RR (complete and partial response)+ of intermittent sunitinib or bevacizumab administered with combination cisplatin and gemcitabine as systemic therapy for locally advanced or metastatic NPC.
  2. To evaluate the pharmacodynamic effects (imaging, circulating and tissue) of intermittent sunitinib or bevacizumab administered with combination cisplatin and gemcitabine as systemic therapy for locally advanced or metastatic NPC.
  3. To evaluate the early pharmacodynamic effects (imaging, circulating and tissue) of 2 loading doses of sunitinib (ie., 12.5mg or 25mg) and 2 dose level of bevacizumab (ie. 7.5mg/kg or 2.5mg/kg) given 1 week prior to administration of cisplatin and gemcitabine chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

Patients may be included in the study only if they meet all of the following criteria:

* Male or female patients aged 21 years and above.
* Patients with histologically confirmed WHO Type II or III NPC.
* Tumour stage III, IVA (T4 N0-2 M0), IVB (Any T N3 M0) or IVC (Any T Any N M1) according to the American Joint Committee on Cancer (AJCC) 2010 criteria. Alternatively, patients with locally advanced recurrent or metastatic NPC for which systemic chemotherapy is indicated will be eligible.
* Eastern Cooperative Oncology Group (ECOG) performance status 0-1.
* Adequate organ function including the following:

  a. Bone marrow function i. Haemoglobin ≥ 9g/dl ii. Absolute neutrophil count (ANC) ≥ 1.5 x 109/L iii. Platelet count ≥ 100 x 109/L.

  b. Liver function i. Bilirubin < or = upper limit of normal (ULN) ii. Alkaline phosphatase (ALP) and gamma-glutamyl transpeptidase (GGT) < or = 2.5x ULN iii. Alanine transaminase (ALT) and aspartate transaminase (AST) < or = ULN iv. Prothrombin time (PT) within the normal range for the institution.

  c. Renal function i. Plasma creatinine within the normal range for the institution or calculated creatinine clearance (by the Cockcroft-Gault formula) > 60mL/min.

  d. Serum amylase and lipase < or = 1.5x ULN.
* Life expectancy of at least 3 months.
* Recovery from any previous drug- or procedure-related toxicity to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE) version 4.0 Grade 0 or 1 (except alopecia), or to baseline preceding the prior treatment.
* Signed informed consent obtained before any study specific procedure. Subjects must be able to understand and be willing to sign the written informed consent.

Exclusion Criteria:

Patients will be excluded from the study for any of the following reasons:

* Previous or concurrent anti-cancer chemotherapy, immunotherapy, radiotherapy or any other investigational therapy.
* Patients who cannot swallow or patients with chronic gastrointestinal disease or conditions that may hamper compliance and/or absorption of the tested product.
* Any concomitant condition that could compromise the objectives of this study and/or the patient's compliance (eg. severe medical conditions such as uncontrolled infection, poorly controlled diabetes mellitus, hypercalcaemia, psychiatric disorders).
* Major thoracic and/or abdominal surgery in the preceding 3 weeks.
* Known human immunodeficiency virus (HIV) seropositivity, hepatitis B or C seropositivity.
* In the investigator's opinion, patients with a current or previous history of clinically significant liver disease within the previous 2 years.
* History of cardiac disease: congestive heart failure > New York Heart Association (NYHA) Class II; active coronary artery disease (unstable angina [anginal symptoms at rest] or new-onset angina [began within the last 3 months] or myocardial infarction within the past 6 months). Cardiac arrhythmias requiring anti-arrhythmic therapy (β-blockers or digoxin are permitted).
* Uncontrolled hypertension (failure of diastolic blood pressure to fall below 90 mmHg, despite the use of ≥ 3 anti-hypertensive drugs or systolic blood pressure greater than 150 mmHg).
* Dehydration NCI-CTCAE Grade 2 or higher.
* Subjects with serious non-healing wound, ulcer, or bone fracture.
* Subjects with arterial or venous thrombotic or embolic events such as cerebrovascular accident (including transient ischemic attacks), deep vein thrombosis, or pulmonary embolism within the 6 months before start of study medication.
* Subjects with renal impairment (creatinine clearance by the Cockcroft-Gault formula) ≤ 60mL/min) or on dialysis.
* Persistent proteinuria of NCI-CTCAE Grade 3 or higher (> 3.5 g/24 hours, measured by urine protein/creatinine ratio on a random urine sample).
* Clinically significant bleeding (NCI-CTCAE Grade 3 or higher) within 30 days prior to start of study medication.
* Subjects unable to swallow oral medications.
* Subjects with seizure disorder requiring anticonvulsant medication.
* History of organ allograft.
* Subjects with evidence or history of disorders of coagulation or thrombosis.
* Pregnancy or breastfeeding.
* Women of childbearing potential not employing adequate contraception. Women of childbearing potential must have a pregnancy test performed a maximum of 7 days before start of study medication, and a negative result must be documented before start of study medication. Women of childbearing potential and men, must agree to use adequate contraception (barrier method of birth control) upon signing the informed consent form until at least 3 months after the last study drug administration. The definition of adequate contraception will be based on the judgment of the treating investigator or a designated associate.
* Substance abuse, medical, psychological or social conditions that may interfere with the subject's participation in the study or evaluation of the study results.
* Known or suspected allergy to the investigational agent or any agent given in association with this study.
* Any condition that is unstable or could jeopardize the safety or compliance of the subject in the study.
* Previous or concurrent cancer which is distinct in primary site or histology from the cancer being evaluated in this study EXCEPT cervical carcinoma in situ, treated basal cell carcinoma, superficial bladder tumors (Ta, Tis & T1) or any cancer curatively treated > 3 years prior to study entry.
* Interstitial lung disease with ongoing signs and symptoms at the time of screening.

Ages: 21 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2011-09-02 (Actual); Primary Completion 2019-03-11 (Actual); Study Completion 2019-03-11 (Actual)

PRIMARY OUTCOMES:
Clinical Response | 2 years
  1. Rates of clinical response (complete and partial clinical response).
  2. Rates of pathological complete responses.
  3. Progression-free survival.
  4. Haematologic and non-haematologic toxicities, as well as serious adverse events.

CONTACTS AND LOCATIONS:
Overall Officials: Boon Cher Goh, MBBS, Principal Investigator — National University Hospital, Singapore
Locations (1):
- National University Hospital, Kent Ridge, Singapore